CLINICAL TRIAL: NCT05704283
Title: 3D Ultrasound Imaging of the Axillary Lymph Nodes
Brief Title: 3D Ultrasound for the Imaging of Lymph Nodes in Patients With Breast Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-006606; NCI-2023-00106 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01EB031040 (NIH)
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Diagnostic (3D-US) (Experimental): Patients undergo 3D-US on study. Patients who have a lymph node clip placed and undergoing neoadjuvant chemotherapy undergo imaging of the clipped node before surgery.
  Interventions: Device: Ultrasound Imaging

INTERVENTIONS:
Device: Ultrasound Imaging — Undergo 3D-US
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US

SUMMARY:
This early phase I studies how well a new 3D ultrasound (3D-US) imaging technology works in evaluating lymph nodes in patients with breast cancer. Ultrasound uses high-frequency sound waves to generate images of the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Conducting a pilot study to optimize the in vivo performance of the newly developed three-dimensional (3D)-ultrasound (US) technology.

II. Evaluate the performance of the new 3D-US technique in differentiating benign from malignant lymph nodes in patients.

III. Compare the performance of the new 3D-US method with conventional two-dimensional (2D)-US for localizing the clipped lymph nodes.

OUTLINE:

Patients undergo 3D-US on study. Patients who have a lymph node clip placed and undergoing neoadjuvant chemotherapy undergo imaging of the clipped node before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lymph node biopsy or lymph node clip placement as per routine clinical care.
* Age of 18 or older.

Exclusion Criteria:

* Vulnerable subjects such as prisoners and adults lacking capacity to consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Lymph node diagnosis by radiologist (benign or malignant) (Aim 2) | Up to 2 years
  Will characterize the lymph node as benign or malignant by reviewing images from each imaging technique based on clinical criteria including node size, shape, margin, cortical thickness, stiffness, and vascularity obtained from B-mode, shear wave elastography, and Doppler imaging. Histopathology results will be used as the ground truth to measure sensitivity and specificity of each ultrasound technology for distinguishing between benign and malignant lymph nodes. The overall agreement of the new 3dimensional (D)-ultrasound (US) method with the biopsy result will be compared to that for 2D-US using McNemar's test. For clipped lymph nodes, the performance of 2D and 3D-US will be compared for localizing the clips.

CONTACTS AND LOCATIONS:
Overall Officials: Shigao D Chen, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials